CLINICAL TRIAL: NCT02701634
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Tolerability of Entospletinib, a Selective SYK Inhibitor, in Combination With Systemic Corticosteroids as First-Line Therapy in Subjects With Chronic Graft Versus Host Disease (cGVHD)
Brief Title: Efficacy and Tolerability of Entospletinib in Combination With Systemic Corticosteroids as First-Line Therapy in Adults With Chronic Graft Versus Host Disease (cGVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-406-1840; 2015-004572-30 (EudraCT Number)
Record Dates: First submitted 2016-02-24; First posted 2016-03-08 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: Chronic Graft Versus Host Disease (cGVHD); newly diagnosed cGVHD; immune reconstitution; Immune System Diseases; allogeneic stem cell transplantation; SYK inhibitor
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Immune System Diseases | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENTO (Experimental): ENTO 400 mg or 200 mg tablet twice daily for 48 weeks
  Interventions: Drug: ENTO
- Placebo (Placebo Comparator): Placebo to match tablet twice daily for 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENTO — Tablets administered orally
  Other Names: GS-9973
  Arms: ENTO
Drug: Placebo — Tablets administered orally
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of entospletinib (ENTO) on the best overall response rate in adults with chronic graft versus host disease (cGVHD) who are currently receiving systemic corticosteroids as part of first-line therapy for cGVHD.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* Male or non-pregnant, non-lactating, females
* Newly diagnosed cGVHD defined by:

  * At least 100 days after receiving any allogeneic hematopoietic stem cell transplant AND
  * Receiving a new course of systemic corticosteroids (≥ 0.5 mg/kg/day) as first-line cGVHD therapy at least 1 day and no more than 21 days prior to first dose of ENTO/Placebo AND
  * Moderate to severe cGVHD as assessed by NIH cGVHD Diagnosis and Staging Criteria (NCDSC) with at least three organ systems involved OR one organ system with a score of 2 OR lung organ score = 1
* Individuals who have undergone transplant for hematologic malignancy are required to be in complete remission.
* Have either a normal ECG or one with abnormalities that are considered clinically insignificant by the investigator in consultation with the Sponsor

Key Exclusion Criteria:

* Inability to begin systemic corticosteroids therapy at a dose of ≥ 0.5 mg/kg/day (or equivalent)
* Uncontrolled infection within 4 weeks prior to randomization
* History of the following therapies in the post-transplant period:

  * B cell depleting biologic agents
  * CD19 CAR-T cells based therapies
  * BTK/SYK/JAK/PI3K inhibitors
  * Phototherapy-unless administered for acute GVHD
* Treatment of cGVHD with anti-thymocyte globulins (ATG), or campath within 60 days of screening visit unless used for treatment of acute GVHD
* Severe organ dysfunction manifested during screening period:

  * Requiring supplemental oxygen at more than 2 L/min
  * Uncontrolled arrhythmia or heart failure

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (30):
- United States (9):
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Taussig Cancer Institute, Cleveland, Ohio
  - Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
- Princess Margaret, Toronto, Ontario, Canada
- France (3):
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint Louis, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum der Universitaet Regensburg, Regensburg
- South Korea (3):
  - Pusan National University Hospital, Busan
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (7):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (3):
  - Kings College Hospital NHS Trust, London
  - St Bartholomew's Hospital, London
  - Manchester Royal Infirmary, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe, Asia, Canada, and United States. The first participant was screened on 27 May 2016. The last study visit occurred on 06 Mar 2018.
Pre-assignment Details: 89 participants were screened.
Groups:
- ENTO: Entospletinib (ENTO) 400 mg or 200 mg tablet twice daily for 48 weeks in combination with systemic corticosteroids as first-line therapy
- Placebo: Placebo to match Entospletinib tablet twice daily for 48 weeks in combination with systemic corticosteroids as first-line therapy
Period: Overall Study
Arm/Group | ENTO | Placebo
Started | 33 | 33
Completed | 1 | 2
Not Completed | 32 | 31
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 0
Not completed — Investigator's Discretion | 7 | 4
Not completed — Study terminated by Sponsor | 15 | 17
Not completed — Withdrew Consent | 6 | 7
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Analysis Set: participants who were randomized into the study. Data was analyzed according to treatment randomized.
Groups:
- ENTO: ENTO 400 mg or 200 mg tablet twice daily for 48 weeks in combination with systemic corticosteroids as first-line therapy
- Placebo: Placebo to match ENTO tablet twice daily for 48 weeks in combination with systemic corticosteroids as first-line therapy
- Total: Total of all reporting groups
Arm/Group | ENTO | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11.9) | 58 (11.4) | 54 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity, Customized: Asian | 3 | 1 | 4
  Race/Ethnicity, Customized: Black | 1 | 0 | 1
  Race/Ethnicity, Customized: White | 23 | 29 | 52
  Race/Ethnicity, Customized: Other | 2 | 0 | 2
  Race/Ethnicity, Customized: Not Permitted | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 21
  Spain | 7 | 10 | 17
  Germany | 5 | 6 | 11
  France | 5 | 3 | 8
  United Kingdom | 3 | 2 | 5
  South Korea | 2 | 1 | 3
  Canada | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: Best overall response rate by 24 weeks was defined as the proportion of participants who achieved a complete or partial overall response as assessed by the NIH cGVHD Activity Assessment (NCAA) within 24 weeks, in the setting of add-on therapy to systemic corticosteroids as part of first-line therapy for cGVHD.
Time Frame: Up to 24 weeks
Population: ITT Analysis Set: all participants who were randomized into the study. Data was analyzed according to treatment randomized.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Placebo to match entospletinib tablets for 48 weeks in combination with systemic corticosteroids as first-line therapy
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 33 | 33
Percentage of participants | 72.7 | 72.7
Statistical Analysis 1: Comparison: ENTO vs Placebo; Test type: Superiority; p = 0.99, Chi-squared — P-value was calculated using the stratified Cochran-Mantel-Haenszel Chi-square test

2. Secondary Outcome: Change From Baseline in the Skin Domain of the Lee Symptom Scale (LSS) at 24 Weeks
Description: The LSS is a patient-reported questionnaire used to measure symptom burden. Each of the LSS subscales ranged between 0 and 100, with higher scores indicating more severe symptoms. A decrease from baseline value correlates with improvement in clinical outcome.
Time Frame: Baseline; Week 24
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale
  Baseline | 15.0 (21.92) | 19.8 (22.34)
  Change at Week 24: number analyzed (Participants) | 9 | 9
  Change at Week 24 | -3.3 (10.31) | -9.4 (14.24)

3. Secondary Outcome: Change From Baseline in the Mouth Domain of the LSS at 24 Weeks
Description: as for outcome 2
Time Frame: Baseline; Week 24
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale
  Baseline | 15.2 (18.17) | 16.8 (21.21)
  Change at Week 24: number analyzed (Participants) | 9 | 9
  Change at Week 24 | -4.2 (16.54) | -1.4 (25.34)

4. Secondary Outcome: Change From Baseline in the Eyes Domain of the LSS at 24 Weeks
Description: as for outcome 2
Time Frame: Baseline; Week 24
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale
  Baseline | 29.4 (27.52) | 21.4 (24.22)
  Change at Week 24: number analyzed (Participants) | 9 | 9
  Change at Week 24 | 10.2 (21.56) | -1.4 (31.32)

5. Secondary Outcome: Change From Baseline in the Total Score of the LSS at 24 Weeks
Description: The LSS is a patient-reported questionnaire used to measure symptom burden. Each of the LSS subscales ranged between 0 and 100, with higher scores indicating more severe symptoms. The total score was calculated by taking the average of the subscale scores. A decrease from baseline value correlates with improvement in clinical outcome.
Time Frame: Baseline; Week 24
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 33 | 33
score on a scale
  Baseline: number analyzed (Participants) | 32 | 32
  Baseline | 16.0 (9.74) | 14.7 (8.51)
  Change at Week 24: number analyzed (Participants) | 9 | 9
  Change at Week 24 | -0.5 (8.35) | -5.4 (8.54)

6. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the documentation of best overall response rate to the documentation of progressive disease. Note that flare was not considered as progressive disease in this analysis.
Time Frame: Up to 48 weeks
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 33 | 33
weeks | 26.3 [9.1 to 44.3] | 32.0 [8.1 to NA] — NA: Not reached
Statistical Analysis 1: Comparison: ENTO vs Placebo; Test type: Superiority; p = 0.67, Log Rank

7. Secondary Outcome: Percentage of Participants Who Achieve at Least 50% Reduction in Systemic Corticosteroid Dose Relative to Baseline
Description: The percentage reduction was calculated as (systemic corticosteroid dose post baseline - baseline systemic corticosteroid dose) / baseline systemic corticosteroid dose.
Time Frame: Baseline; Up to 48 weeks
Population: ITT Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 33 | 33
Percentage of participants | 72.7 | 63.6
Statistical Analysis 1: Comparison: ENTO vs Placebo; Test type: Superiority; p = 0.33, t-test, 2 sided — P-value was calculated using the two sample proportion t-test

8. Secondary Outcome: Percentage of Participants Who Initiate Second-Line Therapy for cGVHD
Description: Second-line therapy for cGVHD was defined as receiving any therapy besides systemic corticosteroids or study drug for the treatment of cGVHD. Inhaled and topical steroids are not considered second-line therapy.
Time Frame: Up to 48 weeks
Population: ITT Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 33 | 33
Percentage of participants | 9.1 | 15.2
Statistical Analysis 1: Comparison: ENTO vs Placebo; Test type: Superiority; p = 0.49, t-test, 2 sided — P-value was calculated using the two sample proportion t-test

9. Secondary Outcome: Failure-Free Survival
Description: Failure-free survival was defined as the time from randomization to the earliest of first documentation of systemic therapy change, nonrelapse mortality, or recurrent malignancy.
Time Frame: Up to 48 weeks
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 20 | 20
Days | 99.0 [57.0 to 214.0] | 85.0 [56.0 to 254.0]
Statistical Analysis 1: Comparison: ENTO vs Placebo; Test type: Superiority; p = 0.800, Log Rank — P-value was calculated using the log-rank test and stratified for disease severity and usage of calcineurin inhibitor or mycophenolate mofetil (MMF); Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.55 to 2.18] — Hazard ratio was estimated from Cox regression model adjusted for treatment and stratified for disease severity and usage of calcineurin inhibitor or MMF

10. Secondary Outcome: Percentage of Participants Who Experience Any Treatment-Emergent Adverse Events (AEs)
Description: Treatment-emergent adverse events are defined as 1 or both of the following: 1) any AEs with an onset on or after study drug or placebo start date and no later than earlier of 30 days after permanent discontinuation of study drug or placebo, 2) any AEs leading to premature discontinuation of study drug or placebo.
Time Frame: Up to 48 weeks plus 30 days
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug, with treatment assignments designated according to actual treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 32 | 33
Percentage of participants | 96.9 | 97.0

11. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 48 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 32 | 33
Percentage of participants | 12.5 | 12.1

12. Secondary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Graded Laboratory Abnormalities
Time Frame: Up to 48 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 32 | 33
Percentage of participants | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (average exposure: ENTO = 18 weeks; Placebo = 17 weeks)
Description: Safety Analysis Set: all participants who received at least 1 dose of study drug, with treatment assignments designated according to actual treatment received.
Arm/Group | ENTO | Placebo
All-Cause Mortality (participants affected / at risk) | 1/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 15/32 | 11/33
Other Adverse Events (participants affected / at risk) | 31/32 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENTO (N=32) | Placebo (N=33)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Disease recurrence (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Listeriosis (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ENTO (N=32) | Placebo (N=33)
Anaemia (Blood and lymphatic system disorders) | 4 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Tachycardia (Cardiac disorders) | 2 | 0
Dry eye (Eye disorders) | 4 | 1
Keratitis (Eye disorders) | 0 | 2
Vision blurred (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Dry mouth (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 4 | 2
Asthenia (General disorders) | 3 | 3
Chest pain (General disorders) | 1 | 2
Fatigue (General disorders) | 8 | 4
Oedema peripheral (General disorders) | 5 | 6
Pyrexia (General disorders) | 5 | 1
Candida infection (Infections and infestations) | 0 | 3
Cytomegalovirus infection (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 2 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
Oral candidiasis (Infections and infestations) | 3 | 1
Respiratory tract infection (Infections and infestations) | 3 | 4
Sinusitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 5
Amylase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 4
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 5 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 0 | 4
Weight increased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Micturition disorder (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Hypertension (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02701634/SAP_000.pdf
  • Study Protocol: Original (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02701634/Prot_001.pdf
  • Study Protocol: Amendment 1 (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02701634/Prot_002.pdf
  • Study Protocol: Amendment 2 (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT02701634/Prot_003.pdf
  • Study Protocol: Amendment 3 (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT02701634/Prot_004.pdf